CLINICAL TRIAL: NCT03813108
Title: Safety and Protective Efficacy of Chemoprophylaxis and Sporozoite Immunization With Plasmodium Falciparum NF135 Against Homologous and Heterologous Challenge Infection in Healthy Volunteers in the Netherlands
Brief Title: Safety and Efficacy of NF135 CPS Immunization
Acronym: CPS135
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject withdrawals after temporal suspension of the trial (for personal, logistic reasons). At time of reinitiation the number of enrolled subjects did not meet the predefined threshold for continuation of the trial.
Sponsor: Radboud University Medical Center (Other)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Principal Investigator, Matthew McCall, dr. MBB McCall, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPS135
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Malaria,Falciparum; Controlled Human Malaria Infection; Immunization; Infection
Keywords: Mosquito bites; Sporozoite; Immunization; Malaria; Falciparum
MeSH Terms: conditions — Malaria, Falciparum; Infections; Malaria | interventions — Mefloquine; Artemether, Lumefantrine Drug Combination; Atovaquone; Proguanil; atovaquone, proguanil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 1: NF135 CPS-immunization challenged by NF135 (Experimental): 10 volunteers will receive three immunizations with 15 NF135.C10 infected Anopheles mosquitoes under mefloquine prophylaxis. Volunteers will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes 19 weeks after the last immunization.
  Interventions: Biological: CPS-immunization; Biological: malaria challenge infection, P. falciparum NF135.C10; Drug: Atovaquone / Proguanil Oral Tablet [Malarone]
- 2: Low dose NF135 CPS-immunization challenged by NF135 (Experimental): 10 volunteers will receive three immunizations with 5 NF135.C10 infected Anopheles mosquitoes under mefloquine prophylaxis. Volunteers will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes 19 weeks after the last immunization.
  Interventions: Biological: CPS-immunization; Biological: malaria challenge infection, P. falciparum NF135.C10; Drug: Atovaquone / Proguanil Oral Tablet [Malarone]
- 3: NF135 CPS-immunization (A/L) challenged by NF135 (Experimental): 10 volunteers will receive three immunizations with 15 NF135.C10 infected Anopheles mosquitoes and are presumptively treated with artemether/lumefantrine starting on day 7 after each immunization. Volunteers will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes.
  Interventions: Biological: malaria challenge infection, P. falciparum NF135.C10; Biological: CPS-immunization (A/L); Drug: Atovaquone / Proguanil Oral Tablet [Malarone]
- 4: NF135 CPS-immunization (A/L) challenged by NF54 (Experimental): 10 volunteers will receive three immunizations with 15 NF135.C10 infected Anopheles mosquitoes and are presumptively treated with artemether/lumefantrine starting on day 7 after each immunization. Volunteers will be challenged by the bites of 5 NF54 infected Anopheles mosquitoes 19 weeks after the last immunization.
  Interventions: Biological: malaria challenge infection, P. falciparum NF54; Biological: CPS-immunization (A/L); Drug: Atovaquone / Proguanil Oral Tablet [Malarone]
- 5: Control group challenged by NF135.C10 Cohort A (Other): Challenge infection control group: 3 volunteers will receive no immunization and will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes 19 weeks after the last immunization.
  Interventions: Biological: malaria challenge infection, P. falciparum NF135.C10; Drug: Atovaquone / Proguanil Oral Tablet [Malarone]
- 6: Control group challenged by NF54 Cohort B (Other): Challenge infection control group: 3 volunteers will receive no immunization and will be challenged by the bites of 5 NF54 infected Anopheles mosquitoes 19 weeks after the last immunization.
  Interventions: Biological: malaria challenge infection, P. falciparum NF54; Drug: Atovaquone / Proguanil Oral Tablet [Malarone]
- 7: Control group challenged by NF135 Cohort B (Other): Challenge infection control group: 3 volunteers will receive no immunization and will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes 19 weeks after the last immunization.
  Interventions: Biological: malaria challenge infection, P. falciparum NF135.C10; Drug: Atovaquone / Proguanil Oral Tablet [Malarone]

INTERVENTIONS:
Biological: CPS-immunization — Subjects will be immunized 3 times by exposure to the bites of P. falciparum NF135.C10 infected mosquitoes while taking mefloquine prophylaxis.
  Other Names: Plasmodium falciparum NF135.C10 sporozoites; Mefloquine
  Arms: 1: NF135 CPS-immunization challenged by NF135; 2: Low dose NF135 CPS-immunization challenged by NF135
Biological: malaria challenge infection, P. falciparum NF135.C10 — Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF135.C10 sporozoites.
  Other Names: Plasmodium falciparum NF135.C10 sporozoites
  Arms: 1: NF135 CPS-immunization challenged by NF135; 2: Low dose NF135 CPS-immunization challenged by NF135; 3: NF135 CPS-immunization (A/L) challenged by NF135; 5: Control group challenged by NF135.C10 Cohort A; 7: Control group challenged by NF135 Cohort B
Biological: malaria challenge infection, P. falciparum NF54 — Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF54 sporozoites.
  Other Names: Plasmodium falciparum NF54 sporozoites
  Arms: 4: NF135 CPS-immunization (A/L) challenged by NF54; 6: Control group challenged by NF54 Cohort B
Biological: CPS-immunization (A/L) — Subjects will be immunized 3 times by exposure to the bites of P. falciparum NF135.C10 infected mosquitoes and receive presumptive treatment with artemether/lumefantrine initiated on day 7 after each immunization.
  Other Names: Plasmodium falciparum NF135.C10 sporozoites; Artemether/lumefantrine (A/L)
  Arms: 3: NF135 CPS-immunization (A/L) challenged by NF135; 4: NF135 CPS-immunization (A/L) challenged by NF54
Drug: Atovaquone / Proguanil Oral Tablet [Malarone] — All participants will be treated with atovaquone/proguanil (1000/400 mg (= 4 tablets) 1×/day during 3 consecutive days) when they develop a malaria infection or on day 28 after malaria challenge infection.

SUMMARY:
This is an open label, randomized, controlled clinical trial. The primary aim of this project is to determine the safety and tolerability of NF135.C10 sporozoite immunization under chemoprophylaxis against homologous and heterologous challenge infection.

DETAILED DESCRIPTION:
A total of 49 healthy volunteers will be allocated to receive either three immunizations with 15 NF135.C10 infected Anopheles mosquitoes (n=30), 3 immunizations with 5 NF135.C10 infected mosquitoes (n=10) or no immunizations (n=6). Immunizations in cohort A (n=20) will be performed under mefloquine prophylaxis, spaced 4 weeks apart. In cohort B, volunteers will not take mefloquine prophylaxis, instead all volunteers will be treated presumptively on day 7 after each immunization with a curative regimen of artemether/lumefantrine, regardless of parasitaemia or symptoms.

Nineteen weeks after the last immunization, all volunteers plus naïve controls will be challenged either by the bites of 5 NF135.C10 (n=36) or 5 NF54 (n=13) infected mosquitoes. After challenge infection, volunteers will be followed up on an out-patient basis once daily for qPCR and safety lab measurements from day 6 until day 21 post challenge. All volunteers will be treated with a curative regimen of atovaquone/proguanil, either at the time of detection of blood stage parasitemia, or 28 days after challenge infection.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 35 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator and is available to attend all study visits.
4. The subject will remain within the Netherlands during the challenge period, not travel to a malaria-endemic area during the study period, and is reachable (24/7) by mobile telephone throughout the entire study period.
5. Subject agrees to inform his/her general practitioner about participation in the study and to sign a request to release by the General Practitioner (GP), and medical specialist when necessary, any relevant medical information concerning possible contra- indications for participation in the study.
6. The subject agrees to refrain from blood donation throughout the study period and for a defined period thereafter according to current guidelines.
7. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study. Acceptable forms of contraception include: established use of oral, injected or implanted hormonal contraceptives; intrauterine device or intrauterine system; barrier methods (condoms or diaphragm with additional spermicide); male partner's sterilisation (with appropriate post-vasectomy documentation of absence of sperm in the ejaculate); true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
8. Subject agrees to refrain from intensive physical exercise (disproportionate to the subjects usual daily activity or exercise routine) during the malaria challenge period.
9. Subject agrees to avoid additional triggers that may cause elevations in liver enzymes including alcohol from baseline up to 1 week post treatment.
10. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following.

   1.1 Body weight <50 kg or Body Mass Index (BMI) <18 or >30 kg/m2 at screening. 1.2 A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiovascular events (including ischemia and myocarditis) in 1st or 2nd degree relatives <50 years old.

   1.3 A medical history of functional asplenia, sickle cell trait/disease, thalassaemia trait/disease or G6PD deficiency.

   1.4 History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   1.5 Screening tests positive for Human Immunodeficiency Virus (HIV), or active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).

   1.6 Chronic use of i) immunosuppressive drugs, ii) antibiotics or antimalarials, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

   1.7 History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.

   1.8 Any history severe psychiatric disease diagnosed by a psychiatrist. 1.9 History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or inclusion, or positive urine toxicology test for cannabis at inclusion.
2. For female subjects: positive urine pregnancy test at screening or at inclusion.
3. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study.
4. Known hypersensitivity to or contra-indications (including co-medication) for use of Mefloquine, Malarone or artemether-lumefantrine, or history of severe (allergic) reactions to mosquito bites.
5. Receipt of any vaccinations in the 3 months prior to the start of the study or plans to receive any other vaccinations during the study period or up to 90 days thereafter.
6. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
7. Being an employee or student of the department of Medical Microbiology of the Radboudumc or the department of Internal Medicine.
8. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew BB McCall, MD PhD DTMH, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] van der Boor SC, Alkema M, van Gemert GJ, Teelen K, van de Vegte-Bolmer M, Walk J, van Crevel R, de Mast Q, Ockenhouse CF, Sauerwein RW, McCall MBB. Whole sporozoite immunization with Plasmodium falciparum strain NF135 in a randomized trial. BMC Med. 2023 Apr 7;21(1):137. doi: 10.1186/s12916-023-02788-9. PMID 37024868

RESULTS

PARTICIPANT FLOW:
Groups:
- 3: NF135 CPS-immunization (A/L) Cohort B: 20 volunteers will receive three immunizations with 15 NF135.C10 infected Anopheles mosquitoes and are presumptively treated with artemether/lumefantrine starting on day 7 after each immunization. Volunteers will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes.
  malaria challenge infection, P. falciparum NF135.C10: 10 Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF135.C10 sporozoites. 10 Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF54 sporozoites.
  CPS-immunization (A/L): Subjects will be immunized 3 times by exposure to the bites of P. falciparum NF135.C10 infected mosquitoes and receive presumptive treatment with artemether/lumefantrine initiated on day 7 after each immunization.
  Atovaquone / Proguanil Oral Tablet [Malarone]: All participants will be treated with atovaquone/proguanil (1000/400 mg (= 4 tablets) 1×/day during 3 consecutive days) when they develop a malaria infection or on day 28 after malaria challenge infection.
Period: Overall Study
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 3: NF135 CPS-immunization (A/L) Cohort B | 5: Control Group Challenged by NF135.C10 Cohort A | 6: Control Group Challenged by NF54 Cohort B | 7: Control Group Challenged by NF135 Cohort B
Started | 10 | 10 | 20 | 3 | 0 | 0
Completed | 8 | 9 | 0 | 3 | 0 | 0
Not Completed | 2 | 1 | 20 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects for groups 6 and 7 were enrolled as the trial was prematurely ended before the challenge infection; control groups were therefore not needed.
Groups:
- 3: NF135 CPS-immunization (A/L) Challenged by NF135 Cohorst B: 20 volunteers will receive three immunizations with 15 NF135.C10 infected Anopheles mosquitoes and are presumptively treated with artemether/lumefantrine starting on day 7 after each immunization. 10 volunteers will be challenged by the bites of 5 NF135.C10 infected Anopheles mosquitoes. 10 volunteers will be challenged by the bites of 5 NF54 infected Anopheles mosquitoes.
  malaria challenge infection, P. falciparum NF135.C10: Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF135.C10 sporozoites.
  CPS-immunization (A/L): Subjects will be immunized 3 times by exposure to the bites of P. falciparum NF135.C10 infected mosquitoes and receive presumptive treatment with artemether/lumefantrine initiated on day 7 after each immunization.
  Atovaquone / Proguanil Oral Tablet [Malarone]: All participants will be treated with atovaquone/proguanil (1000/400 mg (= 4 tablets) 1×/day during 3 consecutive days) when they develop a malaria infection or on day 28 after malaria challenge infection.
- Total: Total of all reporting groups
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 3: NF135 CPS-immunization (A/L) Challenged by NF135 Cohorst B | 5: Control Group Challenged by NF135.C10 Cohort A | 6: Control Group Challenged by NF54 Cohort B | 7: Control Group Challenged by NF135 Cohort B | Total
Number analyzed (Participants) | 10 | 10 | 20 | 3 | 0 | 0 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20 | 3 | 0 | 0 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 24 [20 to 29] | 23.5 [21 to 27] | 23.0 [18 to 30] | 21 [20 to 24] |  |  | 23 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 10 | 2 |  |  | 23
  Male | 3 | 6 | 10 | 1 |  |  | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 7 | 8 | 15 | 3 |  |  | 33
  Race: Asian | 2 | 1 | 0 | 0 |  |  | 3
  Race: Other | 1 | 1 | 5 | 0 |  |  | 7
Region of Enrollment [Number; unit: participants]
  Netherlands | 10 | 10 | 20 | 3 |  |  | 43
Body Mass Index (kg/m^2) [Median (Full Range); unit: kg/m^2] | 23.2 [19.4 to 29.3] | 23.7 [19.8 to 29.7] | 23.4 [18.4 to 29.9] | 22 [21.9 to 23.2] |  |  | 23.2 [18.4 to 29.9]
Hemoglobin (mmol/L) [Median (Full Range); unit: mmol/L] | 9.3 [6.7 to 10.8] | 9.0 [7.6 to 10.1] | 9.0 [7.1 to 9.6] | 8.3 [8.2 to 8.9] |  |  | 9.0 [6.7 to 10.8]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events After NF135.C10 CPS Immunization
Description: The number of adverse events will be recorded by the trial clinicians for all participants.
Time Frame: Cohort A: Inclusion until 35 days after challenge infection (35 weeks) Cohort B: Inclusion - premature end of study (22 weeks)
Population: The Control Group Challenged by NF135.C10 Cohort A, was not included in this analysis as it served only as infection control. As subjects in cohort B did not complete their immunizations they were not yet randomized for infection when the trial ended prematurely. Cohort is therefore analyzed as one group that received 1 immunization with 15 NF135.C10 infected mosquitoes under presumptive A/L treatment.
Measure: Number; unit: Adverse events
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 3: NF135 CPS-immunization (A/L) Cohort B
Number analyzed (Participants) | 10 | 10 | 20
Adverse events | 139 | 173 | 172

2. Primary Outcome: Magnitude of Adverse Events After NF135.C10 CPS Immunization
Description: The severity of adverse events will be recorded (mild/moderate/severe) for each adverse event
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Adverse events
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 3: NF135 CPS-immunization (A/L) Cohort B
Number analyzed (Participants) | 10 | 10 | 20
Adverse events
  Mild adverse events (grade 1) | 108 | 128 | 121
  Moderate adverse events (grade 2) | 20 | 35 | 31
  Severe adverse events (grade 3) | 11 | 10 | 19
  Serious adverse events (grade 4) | 0 | 0 | 1

3. Secondary Outcome: Time to Parasitemia
Description: The effectiveness of CPS-immunization with NF135 sporozoites to protect against malaria challenge infection with homologous N135.C10 or heterologous NF54 sporozoites will be determined by the time to parasitemia in immunized versus non-immunized volunteers after the challenge infection.
Time Frame: Day 1 - 28 after malaria challenge infection (28 days)
Population: The trial was prematurely ended before the challenge infection in cohort B. Only arms that received challenge infection are included in this analysis. In arm 1, 2 subjects withdrew from the trial before challenge infection and 3 subjects were sterily protected and not included in the analysis. In arm 2, 1 subject withdrew from the trial before challenge infection and 2 subjects were sterily protected and not included in this analysis
Measure: Median (Full Range); unit: days to parasitaemia
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 5: Control Group Challenged by NF135.C10 Cohort A
Number analyzed (Participants) | 5 | 7 | 3
days to parasitaemia | 9 [7 to 11] | 7 [7 to 11] | 7 [7 to 7]

4. Post Hoc Outcome: Break Through Infections
Description: Number of subjects that required rescue treatment with atovaquone/proguanil due to a positive thick smear in combination with symptoms following NF135.C10 immunizations despite mefloquine prophylaxis (Cohort A) or presumptive artemether/lumefantrine treatment (Cohort B).
Time Frame: From day 0 until 28 days after each immunization (28 days)
Population: Only study groups that received NF135.C10 immunizations were included in this analysis. One subject in group 2: Low dose NF135 CPS-immunization challenged by NF135, withdrew consent after the first immunization, and thus did not receive immunization 2 and 3. The study was prematurely terminated, therefore subjects in group 3: NF135 CPS-immunization (A/L) Cohort B only received immunization 1.
Measure: Number; unit: participants
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 3: NF135 CPS-immunization (A/L) Cohort B
Number analyzed (Participants) | 10 | 10 | 20
participants
  Break through following immunization 1 | 10 | 10 | 2
  Break through following immunization 2: number analyzed (Participants) | 10 | 9 | 0
  Break through following immunization 2 | 3 | 3 |
  Break through following immunization 3: number analyzed (Participants) | 10 | 9 | 0
  Break through following immunization 3 | 4 | 5 |

ADVERSE EVENTS:
Time Frame: Groups 1 and 2 (Cohort A ): Inclusion until 35 days after challenge infection (35 weeks) Group 3 (Cohort B): Inclusion until premature end of study (22 weeks) Group 5 (Cohort A): Inclusion until 35 days after challenge infection (5 weeks)
Description: As subjects in cohort B did not complete their immunizations, they were not yet randomized for infection when the trial ended prematurely. Cohort B is therefore analyzed as one group that received 1 immunization with 15 NF135.C10 infected mosquitoes under presumptive A/L treatment.
Arm/Group | 1: NF135 CPS-immunization Challenged by NF135 | 2: Low Dose NF135 CPS-immunization Challenged by NF135 | 3: NF135 CPS-immunization (A/L) Cohort B | 5: Control Group Challenged by NF135.C10 Cohort A
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/20 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/20 | 0/3
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 20/20 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: NF135 CPS-immunization Challenged by NF135 (N=10) | 2: Low Dose NF135 CPS-immunization Challenged by NF135 (N=10) | 3: NF135 CPS-immunization (A/L) Cohort B (N=20) | 5: Control Group Challenged by NF135.C10 Cohort A (N=3)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Chest pain, dynamic ECG and elevated cardiac biomarkers 10 days after NF135 immunization. MRI, Coronary CT-A, CAG and echocardiography: no evidence of myocarditis, Tako Tsubo or coronary occlusion/dissection. Inflammatory response most likely.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: NF135 CPS-immunization Challenged by NF135 (N=10) | 2: Low Dose NF135 CPS-immunization Challenged by NF135 (N=10) | 3: NF135 CPS-immunization (A/L) Cohort B (N=20) | 5: Control Group Challenged by NF135.C10 Cohort A (N=3)
Fever (Infections and infestations) | 8 (19) | 8 (16) | 18 (39) | 0 (0)
Chills (Infections and infestations) | 1 (1) | 2 (3) | 9 (13) | 0 (0)
Sweats (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Abdominal pain (Infections and infestations) | 2 (2) | 2 (2) | 3 (4) | 1 (2)
Fatigue (Infections and infestations) | 6 (8) | 5 (12) | 7 (10) | 1 (2)
Headache (Infections and infestations) | 10 (35) | 10 (62) | 18 (37) | 1 (2)
Malaise (Infections and infestations) | 7 (13) | 4 (4) | 12 (16) | 0 (0)
Myalgia (Infections and infestations) | 6 (11) | 6 (20) | 11 (13) | 1 (1)
Nausea (Infections and infestations) | 8 (20) | 8 (17) | 7 (10) | 2 (3)
Decreased appetite (Infections and infestations) | 2 (2) | 1 (1) | 6 (6) | 0 (0)
Dizziness (Infections and infestations) | 1 (1) | 5 (6) | 7 (7) | 0 (0)
Diarrhoea (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Insomnia (General disorders) | 2 (2) | 4 (7) | 0 (0) | 0 (0)
Vivid dreams (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Sadness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
restlessness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Arthralgia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Infections and infestations) | 10 (15) | 7 (10) | 2 (2) | 0 (0)
Erythema (Infections and infestations) | 3 (3) | 1 (3) | 0 (0) | 0 (0)
Swelling (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Canker sores (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
- Early termination of cohort B; heterologous protection could not be assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03813108/Prot_SAP_000.pdf